CLINICAL TRIAL: NCT03687372
Title: A Phase 3 Randomized, Double-Blind, Vehicle-Controlled, Parallel Group Study of A-101 Topical Solution Applied Twice a Week in Subjects With Common Warts
Brief Title: Study of A-101 Topical Solution for the Treatment of Common Warts
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aclaris Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A-101-WART-301
Record Dates: First submitted 2018-09-20; First posted 2018-09-27 (Actual); Results first posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Common Wart
Keywords: common warts
MeSH Terms: conditions — Warts | interventions — N-phenylacetoaminomethylene-DL-p-nitrophenylalanine; 2-Propanol

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Vehicle-Controlled, Parallel Group Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The blinded vehicle solution is packaged to match the active study drug and will be stored under the same conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- A-101 (Experimental): topical solution
  Interventions: Drug: A-101
- Vehicle (Other): topical solution
  Interventions: Other: vehicle

INTERVENTIONS:
Drug: A-101 — hydrogen peroxide topical solution 45%
  Other Names: hydrogen peroxide 45%
  Arms: A-101
Other: vehicle — vehicle as a topical solution
  Other Names: isopropyl alcohol and sterile water
  Arms: Vehicle

SUMMARY:
A Phase 3 Study of A-101 Topical Solution Applied Twice a Week in Subjects with Common Warts

DETAILED DESCRIPTION:
A Phase 3 Randomized, Double-Blind, Vehicle-Controlled, Parallel Group Study of A-101 Topical Solution Applied Twice a Week in Subjects with Common Warts

ELIGIBILITY:
Inclusion Criteria:

1. Subject or legal guardian is able to comprehend and is willing to sign an informed consent/assent for participation in this study.
2. Male or female ≥ 1 years old.
3. Subject has a clinical diagnosis of common warts (verruca vulgaris).
4. Subject has at least 1 and up to 6 clearly identifiable common warts located on the trunk or extremities that meet the requirements as defined below:

   1. Have a longest axis that is ≥3 and ≤8 mm and have a thickness of ≤3mm
   2. Be a discrete lesion, i.e. each wart meeting the entry criteria is clearly separated from other warts.
   3. Be present for at least 4 weeks
   4. Not be covered with hair which, in the investigator's opinion, would interfere with the study medication treatment or the study evaluations
   5. Not be in an intertriginous fold
   6. Periungual, subungual, genital, anal, mosaic, plantar, flat and filiform warts are excluded from treatment and evaluation. If a subject has these types of warts, but also has warts that meet the inclusion criteria, the subject will NOT be excluded from the study.
5. Each common wart identified for treatment must have a PWA ≥ 2.
6. Subject's chemistry and complete blood count results are within normal limits.
7. Subject is in good general health and free of any known disease state or physical condition.
8. Subject is willing and able to follow all study instructions and to attend all study visits.
9. Subject must be the only individual in a household participating in the study.

Exclusion Criteria:

1. Subject has clinically atypical warts.
2. Subject is immunocompromised (e.g., due to chemotherapy, systemic steroids, genetic immunodeficiency, transplant status, etc.).
3. Subject has a history of Human Immunodeficiency Virus (HIV) infection.
4. Subject has had any Human Papilloma Virus (HPV) vaccine within 6 months prior to Visit 1.
5. Subject has used any of the following intralesional therapies within the specified period prior to Visit 2:

   * Immunotherapy (e.g., Candida antigen, mumps antigen, Trichophyton antigen); 8 weeks
   * Anti-metabolite therapy (e.g., bleomycin, 5-fluorouracil); 8 weeks
6. Subject has used any of the following systemic therapies within the specified period prior to Visit 2:

   * Immunomodulatory/immunosuppressant therapy (e.g., etanercept, alefacept, infliximab); 16 weeks
   * Glucocorticosteroids (inhaled and intra-nasal steroids are permitted); 28 days
7. Subject has used any of the following topical therapies within the specified period prior to Visit 2 on, or in the proximity to any of the common warts identified for treatment, that in the investigator's opinion interferes with the study medication treatment or the study assessments:

   * LASER, light or other energy-based therapy (e.g., intense pulsed light [IPL], photodynamic therapy [PDT]); 180 days
   * Immunotherapy (e.g., imiquimod, squaric acid dibutyl ester[SADBE], etc.) 12 weeks
   * Liquid nitrogen, electrodesiccation, curettage; 60 days
   * Hydrogen peroxide; 90 days
   * Antimetabolite therapy (e.g., 5-fluorouracil); 8 weeks
   * Retinoids; 90 days
   * Over-the-counter (OTC) wart therapies and cantharidin; 28 days
8. Subject currently has or has had any of the following within the specified period prior to Visit 1 on or in the proximity to any of the common warts identified for treatment that, in the investigator's opinion, interferes with the study medication treatment or the study assessments:

   * Cutaneous malignancy; 180 days
   * Sunburn; currently
   * Pre-malignancy (e.g., actinic keratosis); currently
9. Subject has a history of sensitivity to any of the ingredients in the study medications.
10. Subject has any current skin or systemic disease (e.g., psoriasis, atopic dermatitis, eczema, sun damage), or condition (e.g., sunburn, excessive hair, open wounds) that, in the opinion of the investigator, might put the subject at undue risk by study participation or interfere with the study conduct or evaluations.
11. Participation in another therapeutic investigational drug/device trial in which administration of an investigational treatment occurred with 30 days prior to Visit 1.
12. Subject has an active malignancy.
13. Subjects is viewed by the Principal Investigator as not being able to complete the study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 503 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-09-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - Aclaris Investigational Site, Mobile, Alabama
  - Aclaris Investigational Site, Hot Springs, Arkansas
  - Aclaris Investigational Site, Fountain Valley, California
  - Aclaris Investigational site, San Diego, California
  - Aclaris Investigational Site, Aventura, Florida
  - Aclaris Investigational Site, Jacksonville, Florida
  - Aclaris Investigational Site, Miami, Florida
  - Aclaris Investigational Site, Ocala, Florida
  - Aclaris Investigational Site, Newnan, Georgia
  - Aclaris Investigational Site, Indianapolis, Indiana
  - Aclaris Investigational Site, Louisville, Kentucky
  - Aclaris Investigational Site, Chestnut Hill, Massachusetts
  - Aclaris Investigational Site, Warren, Michigan
  - Aclaris Investigational Site, Fridley, Minnesota
  - Aclaris Investigational Site, Las Vegas, Nevada
  - Aclaris Investigational Site, Verona, New Jersey
  - Aclaris Investigational Site, Broomall, Pennsylvania
  - Aclaris Investigational Site, Fort Washington, Pennsylvania
  - Aclaris Investigational Site, Charleston, South Carolina
  - Aclaris Investigational Site, Greenville, South Carolina
  - Aclaris Investigational Site, Austin, Texas
  - Aclaris Investigational Site, Pflugerville, Texas
  - Aclaris Investigational Site, San Antonio, Texas
  - Aclaris Investigational Site, Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Hydrogen Peroxide 45% A-101: Topical solution, hydrogen peroxide 45% A-101: hydrogen peroxide 45% topical solution
- Isopropyl Alcohol and Water Vehicle: Topical solution, isopropyl alcohol and water Vehicle: Vehicle solution containing isopropyl alcohol and water
Period: Overall Study
Arm/Group | Hydrogen Peroxide 45% A-101 | Isopropyl Alcohol and Water Vehicle
Started | 254 | 249
Completed | 237 | 210
Not Completed | 17 | 39
Not completed — Lost to Follow-up | 12 | 21
Not completed — Withdrawal by Subject | 4 | 17
Not completed — Investigator Decision | 1 | 1

BASELINE CHARACTERISTICS:
Population: randomized
Groups:
- Active: Topical solution, hydrogen peroxide 45% A-101: hydrogen peroxide 45% topical solution
- Vehicle: Topical solution, isopropyl alcohol and water Vehicle: Vehicle solution containing isopropyl alcohol and water
- Total: Total of all reporting groups
Arm/Group | Active | Vehicle | Total
Number analyzed (Participants) | 254 | 249 | 503
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 92 | 96 | 188
  Between 18 and 65 years | 155 | 148 | 303
  >=65 years | 7 | 5 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.0 (18.21) | 29.4 (18.30) | 30.2 (18.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142 | 137 | 279
  Male | 112 | 112 | 224
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 45 | 72
  Not Hispanic or Latino | 211 | 193 | 404
  Unknown or Not Reported | 16 | 11 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 8 | 4 | 12
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 4 | 4 | 8
  White | 238 | 236 | 474
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 4 | 5
Region of Enrollment [Number; unit: participants]
  United States | 254 | 249 | 503
Fitzpatrick Skin Type [Count of Participants; unit: Participants]
  I - Always Burns | 15 | 10 | 25
  II - Burns Easily | 94 | 79 | 173
  III - Burns Moderately | 92 | 110 | 202
  IV - Burns Minimally | 40 | 41 | 81
  V - Rarely Burns | 11 | 9 | 20
  VI - Never Burns | 2 | 0 | 2
Prior Treatment of any Wart Treated [Count of Participants; unit: Participants]
  Yes | 124 | 118 | 242
  No | 130 | 131 | 261
Total Warts Treated [Count of Participants; unit: Participants]
  1 | 162 | 141 | 303
  2 | 37 | 49 | 86
  3 | 28 | 22 | 50
  4 | 10 | 15 | 25
  5 | 5 | 9 | 14
  6 | 12 | 13 | 25
Time Since First Appearance of Most Recent Wart Treated (Days) [Mean (Standard Deviation); unit: days] | 1306.0 (1852.41) | 1268.2 (1729.51) | 1287.3 (1791.06)
Time since First Appearance of Least Recent Wart Treated (Days) [Mean (Standard Deviation); unit: days] | 1514.3 (2151.39) | 1404.2 (1734.64) | 1459.9 (1955.46)
Longest Axis of "Largest" Wart Treated (mm) [Mean (Standard Deviation); unit: millimeters] | 5.3 (1.54) | 5.1 (1.53) | 5.2 (1.53)
Thickness of "Largest" Wart Treated (mm) [Mean (Standard Deviation); unit: millimeters] | 1.52 (0.743) | 1.51 (0.715) | 1.51 (0.728)

OUTCOME MEASURES:

1. Primary Outcome: The Primary Efficacy Endpoint is the Number of Subjects Whose Identified Common Warts Are Determined to be Clear on the PWA Scale (PWA=0) at Visit 10 (Day 60)
Description: The primary efficacy endpoint is the number of subjects whose identified common warts are determined to be clear on the Physician Wart Assessment (PWA) scale (PWA=0) at Visit 10 (Day 60).
  Efficacy will be assessed using the Physician's Wart Assessment Scale (PWA) which is a 4 point scale. A higher amount of warts cleared represents a better outcome.
Time Frame: Day 60
Population: The study's primary endpoint was to evaluate the amount of patients achieving a clearance of all baseline WARTS. Patients were stratified by the amount of WARTS at Baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrogen Peroxide 45% A-101 | Isopropyl Alcohol and Water Vehicle
Number analyzed (Participants) | 254 | 249
Participants
  Warts at Baseline - All | 40 | 13
  Warts at Baseline - 1: number analyzed (Participants) | 162 | 141
  Warts at Baseline - 1 | 33 | 10
  Warts at Baseline - 2: number analyzed (Participants) | 37 | 49
  Warts at Baseline - 2 | 2 | 1
  Warts at Baseline - 3: number analyzed (Participants) | 28 | 22
  Warts at Baseline - 3 | 2 | 1
  Warts at Baseline - >3: number analyzed (Participants) | 27 | 37
  Warts at Baseline - >3 | 3 | 1
Statistical Analysis 1: Comparison: Hydrogen Peroxide 45% A-101 vs Isopropyl Alcohol and Water Vehicle; A summary of the wart clearance at Visit 10; Test type: Superiority; p = 0.0003, Mixed Models Analysis — P-Value test comparing the Patients Cleared of All Baseline Warts in the Active (A-101 45%) and vehicle groups; Mean Difference (Final Values) = 3.22, 95% CI 2-sided [1.67 to 6.22]

2. Secondary Outcome: Number of Subjects With Complete Clearance of All Treated Common Warts Between Active and Vehicle on the Physician Wart Assessment (PWA) Scale (PWA=0) at Visit 13 (Day 137)
Description: Number of subjects whose identified common warts are determined to be clear on the Physician Wart Assessment (PWA) scale (PWA=0) at Visit 13 (Day 137).
  Efficacy will be assessed using the Physician's Wart Assessment Scale (PWA) which is a 4 point scale. A higher amount of warts cleared represents a better outcome.
Time Frame: Day 137
Population: The secondary efficacy endpoint is the number of subjects whose identified common warts are determined to be clear on the Physician Wart Assessment (PWA) scale (PWA=0) at Visit 13 (Day 137).
  Efficacy will be assessed using the Physician's Wart Assessment Scale (PWA) which is a 4 point scale.
Measure: Count of Participants; unit: Participants
Groups:
- Hydrogen Peroxide 45% A-101: topical solution
  A-101: hydrogen peroxide topical solution 45%
- Isopropyl Alcohol and Water Vehicle: topical solution
  vehicle: vehicle as a topical solution
Arm/Group | Hydrogen Peroxide 45% A-101 | Isopropyl Alcohol and Water Vehicle
Number analyzed (Participants) | 254 | 249
Participants
  Warts at Baseline - All | 57 | 29
  Warts at Baseline - 1: number analyzed (Participants) | 162 | 141
  Warts at Baseline - 1 | 46 | 21
  Warts at Baseline - 2: number analyzed (Participants) | 37 | 49
  Warts at Baseline - 2 | 3 | 1
  Warts at Baseline - 3: number analyzed (Participants) | 28 | 22
  Warts at Baseline - 3 | 3 | 1
  Warts at Baseline - >3: number analyzed (Participants) | 27 | 37
  Warts at Baseline - >3 | 5 | 6
Statistical Analysis 1: Comparison: Hydrogen Peroxide 45% A-101 vs Isopropyl Alcohol and Water Vehicle; Test type: Superiority — P-Value test comparing the Patients Cleared of All Baseline Warts in the Active (A-101 45%) and vehicle groups; p = 0.0024, Mixed Models Analysis; Mean Difference (Final Values) = 2.14, 95% CI 2-sided [1.30 to 3.52]

3. Secondary Outcome: Mean Per-Subject Percent of All Warts That Were Clear on the Physician Wart Assessment (PWA) Scale Between Active and Vehicle That Are Clear (PWA=0) at Visit 13 (Day 137)
Description: Mean Per-Subject Percent of All Warts That Were Clear on the Physician Wart Assessment (PWA) Scale Between Active and Vehicle That Are Clear (PWA=0) at Day 137.
  Clearance of all treated warts will be assessed using the Physician Wart Assessment (PWA) scale which is a four point scale. A higher amount of warts cleared represents a better outcome.
Time Frame: Day 137
Population: Clearance of all treated warts will be assessed using the Physician Wart Assessment (PWA) scale which is a four point scale.
Measure: Mean (Standard Deviation); unit: percentage of all warts cleared
Arm/Group | Hydrogen Peroxide 45% A-101 | Isopropyl Alcohol and Water Vehicle
Number analyzed (Participants) | 254 | 249
percentage of all warts cleared | 28.6 (2.38) | 14.5 (2.40)
Statistical Analysis 1: Comparison: Hydrogen Peroxide 45% A-101 vs Isopropyl Alcohol and Water Vehicle; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney); Odds Ratio (OR) = 14.12, 95% CI 2-sided [7.5 to 20.8]

4. Secondary Outcome: Number of Subjects With a Single Wart at Baseline Whose Wart Was Clear on the PWA Scale Between Active and Vehicle Group (PWA=0) at Visit 10 (Day 60)
Description: Comparison between Active (A-101 45%) and Vehicle of subjects with a single wart at baseline, whose wart is clear (PWA=0) at Day 60.
  Clearance of the single wart at baseline will be assessed using the Physician Wart Assessment (PWA) scale which is a four point scale. A higher amount of warts cleared represents a better outcome.
Time Frame: Day 60
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrogen Peroxide 45% A-101 | Isopropyl Alcohol and Water Vehicle
Number analyzed (Participants) | 162 | 141
Participants | 33 | 10
Statistical Analysis 1: Comparison: Hydrogen Peroxide 45% A-101 vs Isopropyl Alcohol and Water Vehicle; Test type: Superiority; p = 0.0009, Wilcoxon (Mann-Whitney); Odds Ratio (OR) = 3.22, 95% CI 2-sided [1.55 to 6.65]

5. Secondary Outcome: Median Time for Subjects to Achieve Clearance (PWA=0) of All Treated Common Warts
Description: Comparison between Active (A-101 45%) and Vehicle with respect to the median time to achieve onset of clearance (PWA=0) for all treated warts at Day 137.
  Clearance of all treated warts will be assessed using the Physician Wart Assessment (PWA) scale which is a four point scale. A higher amount of warts cleared represents a better outcome.
Time Frame: Day 137
Population: A median was not able to be calculated in the Vehicle group due to an insufficient number of participants with events.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Hydrogen Peroxide 45% A-101 | Isopropyl Alcohol and Water Vehicle
Number analyzed (Participants) | 254 | 249
days | 84 [60.0 to 139.0] | NA [NA to NA] — A median was not able to be calculated in the Vehicle group due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Hydrogen Peroxide 45% A-101 vs Isopropyl Alcohol and Water Vehicle; Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 2.56

ADVERSE EVENTS:
Time Frame: 137 days; Treatment-emergent adverse events (TEAEs) had a start date on or after the date of Visit 2 (study day 1) and treatment-emergent serious adverse events had a start date on or after the date of Visit 1 (Screening). Collection continued through visit 11 (Day 78)
Description: An adverse event (AE) was any untoward medical occurrence in a patient or clinical investigation subject administered a study medication(s) and that did not necessarily have a causal relationship with the study medication.
  Safety summaries by study medication group will include listings by study medication of adverse events incidences within each MedDRA System Organ Class, and changes from pre-application values in vital signs.
Arm/Group | Active | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/254 | 0/249
Serious Adverse Events (participants affected / at risk) | 1/254 | 1/249
Other Adverse Events (participants affected / at risk) | 153/254 | 67/249
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=254) | Vehicle (N=249)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=254) | Vehicle (N=249)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ear Swelling (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 1 (1)
Eye swelling (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Salivary gland enlargement (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Application site discolouration (General disorders) | 1 (1) | 0 (0)
Application site dryness (General disorders) | 2 (2) | 0 (0)
Application site dysaesthesia (General disorders) | 1 (1) | 0 (0)
Application site erosion (General disorders) | 16 (16) | 3 (3)
Application site erythema (General disorders) | 44 (44) | 5 (5)
Application site fissure (General disorders) | 2 (2) | 0 (0)
Application site haemorrhage (General disorders) | 0 (0) | 2 (2)
Application site hypoaesthesia (General disorders) | 0 (0) | 1 (1)
Application site injury (General disorders) | 0 (0) | 2 (2)
Application site irritation (General disorders) | 3 (3) | 0 (0)
Application site oedema (General disorders) | 10 (10) | 0 (0)
Application site pain (General disorders) | 80 (80) | 6 (6)
Application site pallor (General disorders) | 3 (3) | 0 (0)
Application site paraesthesia (General disorders) | 0 (0) | 1 (1)
Application site pruritus (General disorders) | 26 (26) | 6 (6)
Application site reaction (General disorders) | 3 (3) | 0 (0)
Application site scab (General disorders) | 50 (50) | 1 (1)
Application site ulcer (General disorders) | 2 (2) | 0 (0)
Application site vesicles (General disorders) | 3 (3) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Medical device pain (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Allergy to arthropod sting (Immune system disorders) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 2 (2)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 4 (4)
Nasopharyngitis (Infections and infestations) | 8 (8) | 12 (12)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Otitis media acute (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 5 (5)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 6 (6)
Upper respiratory tract infection (Infections and infestations) | 8 (8) | 12 (12)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Burns first degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
Migraine (Nervous system disorders) | 2 (2) | 0 (0)
Sinus headache (Nervous system disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Varicocele (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nail dystrophy (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Onycholysis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Micrographic skin surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (6):
  • Statistical Analysis Plan (2019-06-05): https://cdn.clinicaltrials.gov/large-docs/72/NCT03687372/SAP_000.pdf
  • Informed Consent Form: ICF (ages 12-17) (2018-07-27): https://cdn.clinicaltrials.gov/large-docs/72/NCT03687372/ICF_001.pdf
  • Study Protocol (2019-02-14): https://cdn.clinicaltrials.gov/large-docs/72/NCT03687372/Prot_002.pdf
  • Informed Consent Form: Main ICF (2018-07-27): https://cdn.clinicaltrials.gov/large-docs/72/NCT03687372/ICF_003.pdf
  • Informed Consent Form: ICF (ages 7-11) (2018-07-27): https://cdn.clinicaltrials.gov/large-docs/72/NCT03687372/ICF_004.pdf
  • Informed Consent Form: PCF Photography (2018-10-29): https://cdn.clinicaltrials.gov/large-docs/72/NCT03687372/ICF_005.pdf